CLINICAL TRIAL: NCT06937489
Title: The Effect of the Changes in Cylinder Power and Axis of Toric Soft Contact Lenses on the Visual Quality, Satisfaction and Vision Acceptability in Astigmatic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Tri Rahayu, SpM(K), FIACLE, Ophthalmologist at the Department of Ophthalmology, Faculty of Medicine Universitas Indonesia Cipto Mangunkusumo Hospital, Indonesia, Indonesia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: 20-07-0813; PUTI Saintekes 2020 Grant (Other: The Directorate of Research and Development at the Universitas Indonesia)
Record Dates: First submitted 2025-04-20; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Astigmatism
Keywords: astigmatism; toric contact lens; axis misalignment; visual acuity
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: This study will compare the effect of undercorrection and axis misalignment of toric SCL in mild and moderate astigmatism on visual acuity, contrast sensitivity, visual satisfaction, and vision acceptability.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, the ophthalmologist conducting the eye examinations, and the outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Undercorrection of toric soft contact lens (Experimental): A disposable toric lens investigated in this work is 2-Weeks Acuvue Moist for Astigmatism (2WAMfA), a common hydrogel conventional toric lenses.
  Interventions: Device: Hydrogel conventional toric lenses with undercorrection of 0.5 D; Device: Hydrogel conventional toric lenses with undercorrection of 1.0 D
- Axis misalignment of toric soft contact lens (Active Comparator): A disposable toric lens investigated in this work is 2-Weeks Acuvue Moist for Astigmatism (2WAMfA), a common hydrogel conventional toric lenses.
  Interventions: Device: Hydrogel conventional toric lenses with -10° axis misalignment; Device: Hydrogel conventional toric lenses with +10° axis misalignment

INTERVENTIONS:
Device: Hydrogel conventional toric lenses with -10° axis misalignment — The assessment visits interval is 1 week and completed exactly on day 14 after their first baseline visit. At each assessment visit, three different cylinder power were tested: 1) full cylinder power, 2) under-correction of cylinder power by 0.5 D, and 3) under-correction of cylinder power by 1.0 DC. Axis was also misaligned by -10° and +10° for each cylinder power alteration. The powers and axis assigned to the participants were randomized during every assessment visit. Baseline assessments and treatment allocations were masked to both patients and physician. All assessments were carried out on the day of observation and recorded on the subject evaluation sheet in accordance with the sample data, in which examinations results.
  Arms: Axis misalignment of toric soft contact lens
Device: Hydrogel conventional toric lenses with +10° axis misalignment — The assessment visits interval is 1 week and completed exactly on day 14 after their first baseline visit. At each assessment visit, three different cylinder power were tested: 1) full cylinder power, 2) under-correction of cylinder power by 0.5 D, and 3) under-correction of cylinder power by 1.0 DC. Axis was also misaligned by -10° and +10° for each cylinder power alteration. The powers and axis assigned to the participants were randomized during every assessment visit. Baseline assessments and treatment allocations were masked to both patients and physician. All assessments were carried out on the day of observation and recorded on the subject evaluation sheet in accordance with the sample data, in which examinations results.
  Arms: Axis misalignment of toric soft contact lens
Device: Hydrogel conventional toric lenses with undercorrection of 0.5 D — The assessment visits interval is 1 week and completed exactly on day 14 after their first baseline visit. At each assessment visit, three different cylinder power were tested: 1) full cylinder power, 2) under-correction of cylinder power by 0.5 D, and 3) under-correction of cylinder power by 1.0 DC. Axis was also misaligned by -10° and +10° for each cylinder power alteration. The powers and axis assigned to the participants were randomized during every assessment visit. Baseline assessments and treatment allocations were masked to both patients and physician. All assessments were carried out on the day of observation and recorded on the subject evaluation sheet in accordance with the sample data, in which examinations results.
  Arms: Undercorrection of toric soft contact lens
Device: Hydrogel conventional toric lenses with undercorrection of 1.0 D — The assessment visits interval is 1 week and completed exactly on day 14 after their first baseline visit. At each assessment visit, three different cylinder power were tested: 1) full cylinder power, 2) under-correction of cylinder power by 0.5 D, and 3) under-correction of cylinder power by 1.0 DC. Axis was also misaligned by -10° and +10° for each cylinder power alteration. The powers and axis assigned to the participants were randomized during every assessment visit. Baseline assessments and treatment allocations were masked to both patients and physician. All assessments were carried out on the day of observation and recorded on the subject evaluation sheet in accordance with the sample data, in which examinations results.
  Arms: Undercorrection of toric soft contact lens

SUMMARY:
Toric SCL combined spheric lens power with cylinder power and axis. However, in Indonesia, the availability of cylinder power and axis parameter variations between products are still narrow, with stock-keeping units (SKUs) options only between 0.75-2.75 DC and 10o-180o for power and axis, respectively. Providing accurate toric SCL prescription for astigmatism patient in Indonesia remains a challenge for ophthalmologists and generally could not be achieved. Therefore, the aim of this study is to investigate the effect of power undercorrection and axis misalignment on visual acuity, contrast sensitivity, visual clarity, visual satisfaction, and vision acceptability.

The inclusion criteria for the trial, include: (1) 20 to 40 years of age without the need for presbyopic correction, (2) mild to moderate myopia patients, sphere between -1.00 and - 6.00 D combined with cylinder between -0.75 to -3.00 DC in at least one eye, (3) corrected distance visual acuity (VA) of with Toric SCL 6/15 or better bilaterally. Exclusion criteria include: (1) a history of contact lens use 6 months prior to trial, (2) history of previous ocular surgery, (3) anterior and posterior segment abnormalities, (4) manifest strabismus or dry eye, and (5) ocular and systemic diseases that would preclude CL wear or decrease visual acuity; and pregnancy or lactation.

DETAILED DESCRIPTION:
Detailed Procedure

Baseline refraction and clinical manifestations were determined during initial visit which each participants attended three assessment visits on a separate day. Baseline visual acuity was measured using Snellen chart, contrast sensitivity was measured using Pelli-Robson chart, and VAS (Visual Analog Scale, with 10 being the best indicator) was utilized to measure monocular clarity (1=blurred, 10=clear), satisfaction (1=satisfied, 10=unsatisfied), and vision acceptability (1=unacceptable, 10=perfectly acceptable).

Participants were fitted on their diseased eye, which could be unilateral or bilateral, with the toric SCL. Lens fit (corneal coverage, centration, movement, and rotation) was examined using slit-lamp examination. Regarding lens rotation, modification of the toric SCL axis was determined using the "LARS" (left add, right subtract) method for proper contact lens fitting. The shifting axis in toric SCL was assessed by observing the shift marker on contact lens in a clockwise or anticlockwise direction; then if any, it was corrected using LARS formula. A disposable toric lens investigated in this work is 2-Weeks Acuvue Moist for Astigmatism (2WAMfA), a common hydrogel conventional toric lenses.

The assessment visits interval is 1 week and completed exactly on day 14 after their first baseline visit. At each assessment visit, three different cylinder power were tested: 1) full cylinder power, 2) under-correction of cylinder power by 0.5 D, and 3) under-correction of cylinder power by 1.0 DC. Axis was also misaligned by -10° and +10° for each cylinder power alteration. The powers and axis assigned to the participants were randomized during every assessment visit. Baseline assessments and treatment allocations were masked to both patients and physician. All assessments were carried out on the day of observation and recorded on the subject evaluation sheet in accordance with the sample data, in which examinations results.

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 40 years of age without the need for presbyopic correction
2. mild to moderate myopia patients, sphere between -1.00 and - 6.00 D combined with cylinder between -0.75 to -3.00 DC in at least one eye
3. corrected distance visual acuity (VA) of with Toric SCL 6/15 or better bilaterally.

Exclusion Criteria:

1. a history of contact lens use 6 months prior to trial
2. history of previous ocular surgery
3. anterior and posterior segment abnormalities
4. manifest strabismus or dry eye
5. ocular and systemic diseases that would preclude CL wear or decrease visual acuity; and pregnancy or lactation.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Week 1 and week 2
  Visual acuity was measured using Snellen chart and reported with logMAR
Contrast sensitivity was measured using Pelli-Robson chart, | Week 1 and week 2
  Contrast sensitivity was measured using Pelli-Robson chart,
Monocular clarity | Week 1 and week 2
  VAS (Visual Analog Scale, with 10 being the best indicator) was utilized to measure monocular clarity (1=blurred, 10=clear)
Visual satisfaction | Week 1 and week 2
  VAS (Visual Analog Scale, with 10 being the best indicator) was utilized to measure visual satisfaction (1=satisfied, 10=unsatisfied)
Vision acceptability | Week 1 and week 2
  VAS (Visual Analog Scale, with 10 being the best indicator) was utilized to measure vision acceptability (1=unacceptable, 10=perfectly acceptable).

CONTACTS AND LOCATIONS:
Overall Officials: Tri Rahayu, MD, Principal Investigator — Department of Ophthalmology, Faculty of Medicine Universitas Indonesia Cipto Mangunkusumo Hospital, Indonesia
Locations (1):
- Department of Ophthalmology, Faculty of Medicine Universitas Indonesia Cipto Mangunkusumo Hospital, Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Due to patient privacy and blinding method, IPD will not be shared.